CLINICAL TRIAL: NCT00093587
Title: Pilot Trial of Two Dose Levels of Thymoglobulin® as Part of a Myeloablative-Conditioning for a HLA Identical Matched Related Donor (MRD) Stem Cell Transplant With Cyclosporine (CsA) as Posttransplant Graft vs Host Disease (GvHD) Prophylaxis
Brief Title: Antithymocyte Globulin and Cyclosporine in Preventing Graft-Versus-Host Disease in Patients Undergoing Chemotherapy With or Without Radiation Therapy Followed By Donor Stem Cell Transplant for Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000389241; UCLA-0402009-01; GENZ-SMC-101-1026
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2006-01

CONDITIONS: Graft Versus Host Disease; Leukemia
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Congenital Abnormalities | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor bone marrow transplant or peripheral blood stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and cyclosporine after transplant may stop this from happening.

PURPOSE: This randomized clinical trial is studying how well giving antithymocyte globulin together with cyclosporine works in preventing graft-versus-host disease in patients who are undergoing chemotherapy with or without radiation therapy followed by donor stem cell transplant for acute lymphoblastic leukemia or acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the incidence of acute graft-vs-host disease (GVHD) within the first 100 days after transplantation in patients with acute lymphoblastic leukemia or acute myeloid leukemia treated with a myeloablative conditioning regimen comprising cyclophosphamide (with or without radiotherapy) and low- vs high-dose anti-thymocyte globulin followed by allogeneic HLA-matched related stem cell transplantation and cyclosporine.
* Compare the incidence of serious adverse events within the first 100 days after transplantation in patients treated with these regimens.

Secondary

* Compare 100-day and 6-month survival in patients treated with these regimens.
* Compare the severity of acute GVHD in patients treated with these regimens.
* Compare the incidence of culture-proven infections at 100 days and 6 months after transplantation in patients treated with these regimens.
* Compare the incidence of mucositis, in terms of presence, severity, and duration, in patients treated with these regimens.
* Compare the number of days on opiate drugs within the first 30 days after transplantation in patients treated with these regimens.
* Compare the time to engraftment in patients treated with these regimens.
* Compare the incidence of hospitalization within the first 6 months after transplantation, in terms of length of initial stay, cumulative total days, and number of hospitalizations, in patients treated with these regimens.
* Compare the relapse rate and time to relapse in patients treated with these regimens.
* Compare the incidence and severity of chronic GVHD between 100 days and 6 months after transplantation in patients treated with these regimens.

OUTLINE: This is a pilot, randomized, open-label, multicenter study.

* Conditioning: All patients receive a standard myeloablative-conditioning regimen that contains cyclophosphamide IV over 2 hours per center regimen, typically on days -6 to -3. Patients also undergo total body irradiation OR receive busulfan.
* Graft-versus-host disease (GVHD) prophylaxis (as part of conditioning): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive low-dose anti-thymocyte globulin IV over 4-8 hours on days -3 to -1.
  * Arm II: Patients receive high-dose anti-thymocyte globulin IV over 4-8 hours on days -5 to -1.
* Allogeneic hematopoietic stem cell transplantation: Patients in both arms undergo allogeneic peripheral blood stem cell or bone marrow transplantation on day 0.
* Post-transplantation GVHD prophylaxis: Patients in both arms receive cyclosporine IV over 1-4 hours or orally twice daily beginning on day -1 and continuing until approximately day 60 followed by tapering doses until day 180 in the absence of GVHD.

Patients are followed at 7, 14, 21, 30, 100, and 180 days.

PROJECTED ACCRUAL: A total of 30-60 patients (15-30 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of acute myeloid leukemia (AML) or acute lymphoblastic leukemia

  * In first complete remission or second complete remission
* Secondary AML allowed
* HLA-A, -B, and -DRB1 identical related donor available AND must be fully matched at Class II by high-resolution molecular HLA typing (at least 4 digits)
* Currently receiving a myeloablative conditioning regimen that includes cyclophosphamide

  * All patients from a center should receive the same conditioning regimen throughout the study
  * No fludarabine or other purine analogues (e.g. cladribine or pentostatin) as part of conditioning regimen
* No uncontrolled CNS disease

PATIENT CHARACTERISTICS:

Age

* 18 to 55

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin < 2 mg/dL
* ALT and/or AST ≤ 3 times normal

Renal

* Creatinine < 2.0 mg/dL OR
* Creatinine clearance > 50 mL/min

Cardiovascular

* Ejection fraction > 40%
* No severe cardiac disease

Other

* Negative pregnancy test
* Fertile patients must use effective contraception
* No known contraindication to administration of rabbit anti-thymocyte globulin
* No current drug or alcohol abuse
* No significant medical or psychosocial problem or unstable disease state (including, but not limited to, morbid obesity) that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior or concurrent bone marrow transplantation from a donor who has positive serology for HIV, hepatitis B virus, hepatitis C virus, or syphilis
* No IV immunoglobulin prior to engraftment
* No concurrent ex vivo engineered or processed graft (CD34+ enrichment or T-cell depletion)

Chemotherapy

* See Disease Characteristics
* No prior or concurrent methotrexate for graft-vs-host disease prophylaxis

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior experimental agents
* No other concurrent investigational agents

  * Enrollment in investigational studies (i.e., anti-microbial agents) allowed only for life threatening events or after exhausting other treatment modalities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Gary J. Schiller, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States